CLINICAL TRIAL: NCT05626478
Title: Assessing eFficacy and Safety of DEXTENZA 0.4 mg inseRt in Conjunction With Topical Drop Regimen Treating Pain and inflamMation Following Cataract Surgery Compared to SOC Topical Drop Regimen
Brief Title: Assessing eFficacy and Safety of DEXTENZA 0.4 mg inseRt, Following Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nicole Fram M.D. (Other)
Responsible Party: Sponsor-Investigator, Nicole Fram M.D., CEO, Advanced Vision Care
Organization: Advanced Vision Care (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVC-003
Record Dates: First submitted 2022-11-08; First posted 2022-11-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Corneal Edema; Corneal Defect; Anterior Chamber Inflammation; Ocular Pain; Corneal Staining; Visual Outcome; CME - Cystoid Macular Edema
MeSH Terms: conditions — Corneal Edema; Eye Pain; Macular Edema | interventions — Calcium Dobesilate; Dexamethasone; prednisolone acetate; bromfenac; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: In patient who undergo cataract surgery, subjects will be randomized to 2 arms and be followed for a period of 3 months.
  Arm 1- control group, 25 subjects will receive Prednisolone Acetate 1% QID x 2 weeks then BID x 2 weeks.
  Arm 2 - study group, 25 subjects will receive Dextenza 0.4mg insert
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 - Cataract surgery gtt regimen per SOC (Active Comparator): Following cataract surgery (without Dextenza 0.4mg insert) patients will receive: Prednisolone Acetate 1% QID X 2 Weeks, then BID x 2 weeks and stop / Prolensa 0.07% QD X 4 Weeks and stop.
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp; Drug: Prolensa 0.07% Ophthalmic Solution
- Arm 2 - Cataract surgery with Dextenza and less frequency of gtt regimen (Experimental): Following cataract surgery with DEXTENZA 0.4mg insert, patients will receive: Prolensa 0.07% QD X 4 Weeks and stop
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert; Drug: Prolensa 0.07% Ophthalmic Solution

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — DEXTENZA 0.4Mg Ophthalmic Insert is a corticosteroid (to decrease inflammation) intracanalicular insert placed in the punctum, a natural opening in the eye lid, and into the canaliculus and is designed to deliver dexamethasone to the ocular surface for up to 30 days without preservatives.
  Other Names: Dexamethasone 0.4mg
  Arms: Arm 2 - Cataract surgery with Dextenza and less frequency of gtt regimen
Drug: Prednisolone Acetate 1% Oph Susp — Prednisolone Acetate 1% is a corticosteroid (to decrease inflammation) and being used as a topical drop after cataract surgery per Standard Of Care.
  Arms: Arm 1 - Cataract surgery gtt regimen per SOC
Drug: Prolensa 0.07% Ophthalmic Solution — Prolensa 0.07% is a NSAID (to decrease inflammation, swelling and pain) and is being used as a topical drop after cataract surgery per Standard Of Care.

SUMMARY:
Assessing eFficacy and Safety of DEXTENZA 0.4 mg inseRt, Following Cataract Surgery

DETAILED DESCRIPTION:
Assessing eFficacy and Safety of DEXTENZA 0.4 mg inseRt Treating Pain, and inflamMation Following Cataract Surgery Compared to Topical Prednisolone Acetate 1%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clinically significant cataract and are planning to undergo non-complicated Clear Cornea Incision Cataract Extraction with Posterior Capsule IntraOcular Lens in one or both eyes
* Are willing and able to comply with clinic visits and study related procedures
* Are willing and able to sign the informed consent form

Exclusion Criteria:

* Under the age of 18 at the time of signing the Informed Consent Form
* Pregnant or planning to become pregnant during the trial period
* Have visual acuity potential of less than 20/30 as recorded by a Retinal Acuity Meter or Potential Acuity Meter glare testing
* Have active infectious systemic disease
* Have active infectious ocular or extraocular disease
* Have punctal plug in the study eye
* Have obstructed nasolacrimal duct in the study eye(s) (dacryocystitus)
* Have known hypersensitivity to dexamethasone or are a known steroid responder
* Have a history of ocular inflammation or macular edema
* Has history of Laser Vision Correction (LASIK, PhotoRefractive Keratectomy) in the operated eye
* Are currently being treated with immunomodulating agents in the study eye
* Are currently being treated with immunosuppressants and/or oral steroids
* Are currently being treated with corticosteroid implant (i.e Ozurdex)
* Have a history of herpes simplex virus keratitis or present active bacterial, viral, or fungal keratitis in either eye
* Have a history of complete punctal occlusion in one or both punctum
* Currently using topical ophthalmic steroid medications
* Are unwilling or unable to comply with the study protocol
* Are determined by the Investigator to not be included for reasons not already specified (e.g., systemic, behavioral, or other ocular disease/abnormality) if the health of the subject or the validity of the study outcomes may be compromised by the subject's enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Mean change in anterior chamber inflammation (Cell and Flare) scores | Assessed on Days 1,7,30,90
  Measured by SUN (Standardization on Uveitis Nomenclature) grading scale: absence of cell to be defined as a grade of 0-0.5 and absence of flare to be defined as a grade of: 0-1. 0-4 score scale, higher scores mean a worse outcome. 0-1 Absent, 1-2 Mild, 2-3 Moderate, 4 Severe.
Mean change in pain score | Assessed on Day 1,7, 30 and 90
  Measured with the visual analog scale (VAS); between 0 and 100; 0 meaning no pain and 100 meaning worst pain possible, higher scores mean a worse outcome. 0-10 Absent, 11-30 Mild, 31-70 Moderate, 71-100 Severe.

SECONDARY OUTCOMES:
Visual outcome (Best Corrected Visual Acuity) | Assessed on Day 1,7, 30 and 90
  Measured by ETDRS (Early Treatment Diabetic Retinopathy Study) chart. 0-70 letter read score, higher scores mean a better outcome.
Absence of CME (Cystoid Macular Edema) | Assessed on Day 90
  Macular thickness measured by OCT (Optical Coherence Tomography) and compared to the preop measurements, higher scores (>over 50 microns) mean a worse outcome.
Mean change in corneal staining | Assessed on Day 7, 30 and 90
  measured by the National Eye Institute 0-4 score scale, higher scores mean a worse outcome. 0-1 Mild, 2-3 Moderate, 4 Severe. Total score 0-5 Mild, 6-15 Moderate, 16-20 Severe.

OTHER OUTCOMES:
Safety endpoint: corneal or retinal edema | Assessed throughout 90-day study period
  Measured by slit lamp examination and supporting imaging and testing such as Pachymetry measured in micrometer (μm) or Macular OCT (Optical Coherence Tomography) measured in microns (μ). Higher scores (in comparison to preop measurements) mean a worse outcome.
Safety endpoint: Signs of Rebound Iritis | Assessed throughout 90-day study period
  Measured by slit lamp examination and scored by SUN (Standardization on Uveitis Nomenclature) grading scale of Anterior chamber Cell and Flare presence. 0-4 score scale. Cell: 0-0.5 Absence, 1-2 Mild, 2-3 Moderate 4 Severe. Flare: 0-1 Absence, 2 Mild, 3 Moderate, 4 Severe. Higher scores mean a worse outcome. (specifically sub-grouped Blue vs. Brown eyed subjects)
Safety endpoint: Change in IOP (IntraOcular Pressure) initiating rescue medications | Assessed throughout 90-day study period
  Measured by Applanation in millimeter Hg(Mercury), higher then 22mm Hg or lower then 10mm Hg mean a worse outcome and a need for rescue.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Fram, M.D., Principal Investigator — Advanced Vision Care
Locations (1):
- Advanced Vision Care, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenwood MD, Gorham RA, Boever KR. A Randomized Fellow-Eye Clinical Trial to Evaluate Patient Preference for Dexamethasone Intracanalicular Insert or Topical Prednisolone Acetate for Control of Postoperative Symptoms Following Bilateral Femtosecond Laser in Site Keratomileusis (LASIK). Clin Ophthalmol. 2020 Aug 6;14:2223-2228. doi: 10.2147/OPTH.S265311. eCollection 2020. PMID 32821083
- [Background] Tyson SL, Bafna S, Gira JP, Goldberg DF, Jones JJ, Jones MP, Kim JK, Martel JM, Nordlund ML, Piovanetti-Perez IK, Singh IP, Metzinger JL, Mulani D, Sane S, Talamo JH, Goldstein MH; Dextenza Study Group. Multicenter randomized phase 3 study of a sustained-release intracanalicular dexamethasone insert for treatment of ocular inflammation and pain after cataract surgery. J Cataract Refract Surg. 2019 Feb;45(2):204-212. doi: 10.1016/j.jcrs.2018.09.023. Epub 2018 Oct 24. PMID 30367938
- See also: Dextenza [package insert]. Bedford, MA: Ocular Therapeutix, Inc; 2019 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/208742s001lbl.pdf